CLINICAL TRIAL: NCT02142296
Title: A 12-month, Exploratory Open-label Study of Eylea (Aflibercept) in Subjects With Retinal Pigment Epithelial Detachment Secondary to Neovascular Age-related Macular Degeneration
Brief Title: Eylea to Treat Retinal Pigment Epithelial Detachment (RPED) Secondary to Wet Age-Related Macular Degeneration (wAMD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, John Gonder, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bayer-001-PED
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Retinal Pigment Epithelial Detachment Secondary to Age-related Macular Degeneration
Keywords: Pigment Epithelial Detachment; Age-related Macular degeneration
MeSH Terms: conditions — Retinal Detachment; Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eylea (Other): The intravitreal dose of Eylea will be 2mg (50ul) per injection. The medication will be supplied in single use vials. Given monthly for 3 months and then every 8 weeks until week 52. This is an open-label study.
  Interventions: Drug: Eylea

INTERVENTIONS:
Drug: Eylea — monthly injections for 3 months and then every other month to 1 year. volume administered is 0.05ml
  Other Names: Eylea is the brand name.; Aflibercept is the generic name.; The DIN is 02415992.

SUMMARY:
Primary Objectives:

To assess the efficacy of intravitreal administered Eylea in preventing visual loss in subjects with a retinal pigment epithelial detachment (PED) subtype of neovascular age-related macular degeneration (AMD) measured by mean change in BCVA at Month 12 compared to Baseline.

Secondary Objectives:

1. To assess the safety and tolerability of repeated intravitreal administration of Eylea in subjects with the PED subtype of neovascular AMD for a period of 1 year
2. To assess the effect of repeated intravitreal administration of Eylea on Central Subfield Thickness (CSFT), Central Subfield Volume (CSFV), and PED height and volume.
3. To assess the effect of repeated intravitreal administration of Eylea on vision related quality of life in subjects with PED study type of neovascular AMD assessed using the NEI/VFQ-25 questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent.
2. Men and women greater than or equal to 55 years of age.
3. Recent development of RPED secondary to AMD.
4. ETDRS best corrected visual acuities of 20/40 to 20/320 (letter score of 73 to 25) in the study eye.
5. Willing and committed and able to return for all clinic visits and complete all study related procedures.

Exclusion Criteria:

1. Any prior treatment for neovascular AMD except dietary supplements or vitamins. (for patients in the treatment naïve group only)
2. Any prior or concomitant therapy with another investigational agent to treat neovascular AMD in the study eye.
3. Total lesion size greater than 12 disc areas.
4. Subretinal hemorrhage that is either 50% or more of the total lesion area or if the blood is under the fovea and is 1 or more disc areas in size in the study eye.
5. Scar or fibrosis making up greater than 50% of the total lesion in the study eye.
6. Scar, fibrosis or atrophy involving the center of the fovea.
7. Presence of a retinal pigment epithelial tear.
8. History of a vitreous hemorrhage within 4 weeks prior to initiation of the study.
9. Presence of other causes of choroidal neovascular membrane other than AMD.
10. History of clinical evidence of diabetic retinopathy, especially diabetic maculopathy or macular edema from other causes, including retinal vein occlusion or diabetes
11. Prior vitrectomy surgery in the study eye.
12. History of retinal detachment treatment in the study eye.
13. History of macular hole in the study eye.
14. Any intraocular/periocular surgery within 3 months of the initiation of the study.
15. Prior trabeculectomy or filtering surgery in the study eye.
16. Uncontrolled glaucoma, defined as a pressure greater than 25 mmHg despite treatment.
17. Active intraocular inflammation.
18. Active ocular/periocular infection.
19. Any history of uveitis.
20. Active scleritis or episcleritis.
21. Aphakia or pseudophakia with absence of posterior capsule (unless it occurred as a result of YAG posterior capsulotomy) in the study eye.
22. Previous radiation therapy in the region of the study eye.
23. History of corneal transplant or corneal dystrophy in the study eye.
24. Significant medial opacities including cataract that may interfere with visual acuity or fundus photography.
25. Any disease or ocular condition which, in the opinion of the investigator could either increase in the risk to the subject beyond what is expected from a standard procedure of intraocular injections or which may be considered contraindicated for the use of the investigational drug (VEGF Trap).
26. The use of long acting steroids systemically or intraocularly.
27. Any history of allergy to Proviodine or fluorescein sodium.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
efficacy of Eylea in patients with RPED | baseline to month 12
  visual acuity mean change from baseline compared to month 12

SECONDARY OUTCOMES:
safety and tolerability of repeated Eylea injection | period of 1 year
  assessment of adverse events at each visit
effect of repeated Eylea injections of Central Subfield Thickness , Central Subfield Volume and PED height and volume | baseline to month 12
  using OCT (optical coherence tomography) thickness, volume and height will be compared from baseline to month 12
effect of repeated Eyle injections on vision related quality of life | baseline to month 12
  using the standardized NEI/VFQ-25 questionnaire reponses will be compared from baseline to month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Ivey Eye Institute, London, Ontario, Canada

REFERENCES:
- [Derived] Diaconita V, Li B, Pal L, Bahnacy F, Gonder JR. Prospective evaluation of aflibercept in pigment epithelial detachments secondary to neovascular age related macular degeneration. Can J Ophthalmol. 2019 Oct;54(5):626-634. doi: 10.1016/j.jcjo.2019.01.004. Epub 2019 Apr 3. PMID 31564356